CLINICAL TRIAL: NCT07262463
Title: The Effect of Traction-Pressure-Release (TPR) and Manual Pressure Methods on Intramuscular Injection Pain and Satisfaction in Adults: A Randomized Controlled Trial
Brief Title: Effect of Traction-Pressure-Release and Manual Pressure on Intramuscular Injection Pain
Acronym: IM-PainTech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melek Sahin (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Sponsor-Investigator, Melek Sahin, Assistant Professor, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-60116787-020-612652
Record Dates: First submitted 2025-11-20; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Intramuscular Injection Pain
Keywords: Intramuscular injection; Pain; Manual pressure; TPR technique; Ventrogluteal site
MeSH Terms: conditions — Pain | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group, single-blind randomized controlled design with three independent arms. Participants are randomly assigned in a 1:1:1 ratio to one of the following groups: (1) Standard intramuscular injection (control), (2) Manual Pressure technique, or (3) Traction-Pressure-Release (TPR) technique. Each participant receives only one type of intervention, and no crossover or repeated interventions are applied. Outcomes (pain intensity and injection satisfaction) are measured immediately after the injection using validated visual scales. Randomization is performed using block randomization to ensure balance among groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Intramuscular Injection (Control Group) (Other): Control Group: Participants in this arm will receive the standard intramuscular (IM) injection technique without any additional intervention. The injection will be administered into the ventrogluteal site using a 5 mL syringe with a 21G, 38 mm needle. The injection area will be cleaned with an alcohol swab, and the medication (diclofenac sodium, 3 mL) will be delivered at a rate of 1 mL per 10 seconds. No manual pressure or Traction-Pressure-Release (TPR) technique will be applied. Pain and satisfaction will be assessed immediately after the injection using validated visual scales.
  Interventions: Other: Standard Intramuscular Injection
- Manual Pressure Technique (Experimental): Manual Pressure Group: Participants in this arm will receive the intramuscular (IM) injection using the Manual Pressure technique. Before needle insertion, the non-dominant thumb will apply firm pressure to the identified ventrogluteal injection site for 10 seconds. Following skin cleaning with an alcohol swab, diclofenac sodium (3 mL) will be injected at a rate of 1 mL per 10 seconds using a 5 mL syringe with a 21G, 38 mm needle. No traction or rapid muscle release will be applied. Pain and satisfaction will be assessed immediately after the injection using validated visual scales.
  Interventions: Procedure: Manual Pressure Technique
- Traction-Pressure-Release (TPR) Technique (Experimental): TPR Group: Participants in this arm will receive the intramuscular (IM) injection using the Traction-Pressure-Release (TPR) technique. After skin cleaning, the syringe is held in the dominant hand. As the needle is inserted at a 90-degree angle, the non-dominant hand simultaneously applies skin traction with deep pressure, followed by rapid muscle release. After aspiration, diclofenac sodium (3 mL) is injected at a rate of 1 mL per 10 seconds using a 21G, 38 mm needle. The dominant hand remains stable throughout. Pain and satisfaction will be measured immediately after the injection using validated visual scales.
  Interventions: Procedure: Traction-Pressure-Release (TPR) Technique

INTERVENTIONS:
Other: Standard Intramuscular Injection — Participants in this arm will receive the standard intramuscular (IM) injection technique without any additional intervention. The IM injection will be administered into the ventrogluteal site using a 5 mL syringe with a 21G, 38 mm needle. The injection area will be cleaned with an alcohol swab, and diclofenac sodium (3 mL) will be injected at a rate of 1 mL per 10 seconds. No manual pressure or Traction-Pressure-Release (TPR) technique is applied. Pain and satisfaction are assessed immediately after the injection using validated visual scales.
  Arms: Standard Intramuscular Injection (Control Group)
Procedure: Manual Pressure Technique — In this intervention, firm manual pressure is applied to the ventrogluteal injection site using the non-dominant thumb for 10 seconds prior to needle insertion. After cleaning the skin with an alcohol swab, diclofenac sodium (3 mL) is injected at a rate of 1 mL per 10 seconds using a 5 mL syringe with a 21G, 38 mm needle. No traction or rapid muscle release is performed. Pain and satisfaction are measured immediately after the injection using validated visual scales.
  Arms: Manual Pressure Technique
Procedure: Traction-Pressure-Release (TPR) Technique — In this intervention, the IM injection is administered using the Traction-Pressure-Release (TPR) technique. After preparing the site with an alcohol swab, the needle is inserted at a 90-degree angle while the non-dominant hand applies simultaneous skin traction and deep pressure to the injection site. Immediately after needle insertion, the muscle is rapidly released, followed by aspiration and injection of diclofenac sodium (3 mL) at a rate of 1 mL per 10 seconds. The dominant hand holding the syringe remains stable throughout the procedure. Pain and satisfaction are assessed immediately after the injection using validated visual scales.
  Arms: Traction-Pressure-Release (TPR) Technique

SUMMARY:
The goal of this clinical trial is to evaluate whether two different intramuscular (IM) injection techniques-Manual Pressure and Traction-Pressure-Release (TPR)-can effectively reduce injection-related pain and improve patient satisfaction in adult hospitalized patients receiving diclofenac sodium (3 mL) via IM injection.

The main questions the study aims to answer are:

Does the TPR technique reduce IM injection pain more effectively than the standard method?

Does the Manual Pressure technique reduce IM injection pain more effectively than the standard method?

How are patients' fear of injection and experienced pain related?

Since there is a comparison group, researchers will compare three arms (Control, Manual Pressure, TPR) to determine whether either technique results in lower pain scores and higher satisfaction compared with the standard IM injection procedure.

Participants will:

Receive diclofenac sodium via IM injection in the ventrogluteal site using one of three randomized techniques:

* Standard IM injection (Control)
* Manual Pressure technique
* Traction-Pressure-Release (TPR) technique

Rate their pain using the Visual Analog Scale (VAS) immediately after the injection.

Rate their satisfaction using the Injection Satisfaction Scale.

Provide demographic and clinical data through a Patient Information Form.

This study uses a single-blind randomized controlled trial design with three parallel groups. A total of 174 adult patients will be enrolled to ensure adequate power for statistical comparison.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years.

* Hospitalized in the Orthopedics, General Surgery, or Orthopedics Clinic at Servergazi State Hospital.
* Prescribed intramuscular diclofenac sodium (3 mL).
* Has not received any intramuscular injection in the previous week.
* Able to understand instructions and accurately use the Visual Analog Scale (VAS).
* Provides written informed consent.

Exclusion Criteria:

* Presence of pain, abscess, infection, tissue necrosis, hematoma, or any complication related to previous intramuscular injections at the ventrogluteal site.
* Impaired consciousness or communication difficulties.
* Visual or hearing impairment that prevents accurate scale assessment.
* Any physical condition preventing proper positioning of the extremities for IM injection.
* Declines to participate or withdraws consent at any time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity after intramuscular injection | Immediately after injection (within 1-2 minutes)
  Pain intensity will be measured using the 100-mm Visual Analog Scale (VAS), where 0 indicates "no pain" and 100 indicates "worst imaginable pain." Participants will mark their pain level immediately after the intramuscular injection. The distance (mm) from the left end of the scale to the participant's mark will be recorded as the pain score.

SECONDARY OUTCOMES:
Injection satisfaction level | Immediately after injection (within 1-2 minutes)
  Satisfaction will be measured using a 100-mm Visual Satisfaction Scale, where 0 indicates "very dissatisfied" and 100 indicates "very satisfied." Participants will mark their satisfaction immediately after the injection.
Relationship between fear of injection and experienced pain | Immediately after injection
  Participants' reported history of injection fear (Yes/No), recorded on the Patient Information Form, will be analyzed in relation to post-injection VAS pain scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Sıtkı Koçman University, Fethiye Faculty Of Health Sciences, Department of Nursing, Muğla, Fethiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy concerns and institutional policies. Only summary results will be made available.

REFERENCES:
- [Result] Sanlialp Zeyrek A, Takmak S, Kurban NK, Arslan S. Systematic review and meta-analysis: Physical-procedural interventions used to reduce pain during intramuscular injections in adults. J Adv Nurs. 2019 Dec;75(12):3346-3361. doi: 10.1111/jan.14183. Epub 2019 Sep 13. PMID 31452229
- [Result] Cmc S, Lord H, Vargese SS, Kurian N, Cherian SA, Mathew E, Fernandez R. Effectiveness of physical stimulation for reducing injection pain in adults receiving intramuscular injections: a systematic review and meta-analysis. JBI Evid Synth. 2023 Feb 1;21(2):373-400. doi: 10.11124/JBIES-20-00590. PMID 36758552
- [Result] Ozturk D, Baykara ZG, Karadag A, Eyikara E. The effect of the application of manual pressure before the administration of intramuscular injections on students' perceptions of postinjection pain: a semi-experimental study. J Clin Nurs. 2017 Jun;26(11-12):1632-1638. doi: 10.1111/jocn.13530. Epub 2016 Nov 24. PMID 27535654
- [Result] Salari M, Estaji Z, Akrami R, Rad M. Comparison of skin traction, pressure, and rapid muscle release with conventional method on intramuscular injection pain: A randomized clinical trial. J Educ Health Promot. 2018 Dec 28;7:172. doi: 10.4103/jehp.jehp_216_18. eCollection 2018. PMID 30693308